CLINICAL TRIAL: NCT01979159
Title: A Novel Treatment for Aphasia and Apraxia of Speech: Measurement of Outcomes
Brief Title: A Novel Treatment for Aphasia and Apraxia of Speech : Measurement of Outcomes
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: VA Office of Research and Development (U.S. Federal Agency)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: O1356-P
Record Dates: First submitted 2013-10-23; First posted 2013-11-08 (Estimated); Results first posted 2019-06-19 (Actual); Last update posted 2019-06-19 (Actual); Status verified 2019-03

CONDITIONS: Apraxia of Speech; Aphasia
Keywords: aphasia; apraxia of speech; outcomes
MeSH Terms: conditions — Apraxias; Aphasia

STUDY DESIGN:
Intervention Model Description: Single-case experimental design; multiple baseline design across behaviors and participants
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (1):
- Combined Aphasia-ApraxiaTreatment (Experimental): Administration of Combined Aphasia and Apraxia of Speech Treatment )(CAAST) to 4 persons with aphasia and apraxia of speech in the context of single-subject designs
  Interventions: Behavioral: Combined Aphasia and Apraxia of Speech Treatment (CAAST)

INTERVENTIONS:
Behavioral: Combined Aphasia and Apraxia of Speech Treatment (CAAST) — Therapy is delivered in a face-to-face format. The therapist uses picture stimuli, verbal modeling, feedback, reinforcement, forward-chaining to increase verbal production. For speech errors that occur, the therapist uses modeling, feedback, reinforcement, simultaneous production, articulatory instruction, and repeated practice to improve articulation.
  Other Names: CAAST

SUMMARY:
In order to determine if speech-language therapy has positive effect, reliable measurement tools are required to document outcomes. Currently, there is very limited information concerning the measurement of changes in speech production as a result of treatment for acquired apraxia of speech and aphasia. This study will obtain information concerning the reliability of several speech production measures over time. Thirty persons with chronic aphasia and apraxia of speech will be asked to provide speech samples in response to commonly used assessment tools on three sampling occasions so that the stability of measurements may be examined.

After establishment of appropriate outcome measures, a small, pilot treatment study will be conducted with four participants. The participants will receive a new treatment for aphasia and acquired apraxia of speech and outcomes will be measured relative to speech and language production.

DETAILED DESCRIPTION:
A single group, repeated measures design will be used to obtain repeated speech samples from 30 persons with chronic acquired apraxia of speech and aphasia. Speech samples will be elicited using commonly employed motor speech assessment protocols; an initial sample, a sample one week following the initial sample, and a sample at four weeks following the initial sample. The following measures will be obtained from the samples: percent consonants correct, percent fluent utterances, and duration of utterance. Stability of the measures will be examined.

After the preceding measures have been analyzed, a series of four, single-subject experimental designs will be conducted. Four participants with chronic aphasia and apraxia of speech will receive a new treatment for aphasia and apraxia of speech applied sequentially to two sets of experimental picture picture stimuli. Outcomes will be measured in terms of speech production (measures described above) as well as in terms of language production.

ELIGIBILITY:
Inclusion Criteria:

* Veterans or non Veterans with aphasia and apraxia of speech who reside in the Salt Lake City region (commutable),
* 12 months or more post stroke or other focal brain injury, no other neurological conditions,
* native English speakers, hearing adequate for experimental task (e.g., pass puretone screening at 35dB at 500, 1K, 2K Hz),
* non linguistic cognition within normal limits

Exclusion Criteria:

* less than 12 months post stroke,
* insufficient hearing, insufficient non linguistic cognitive skills,
* neurological conditions other than stroke,
* more than one stroke or brain injury
* unable to attend treatment in the Salt Lake City vicinity

Ages: 21 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 4 (Actual)
Dates: Start 2013-10-21 (Actual); Primary Completion 2016-12-30 (Actual); Study Completion 2017-12-22 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Julie L Wambaugh, PhD, Principal Investigator — VA Salt Lake City Health Care System, Salt Lake City, UT
Locations (1):
- VA Salt Lake City Health Care System, Salt Lake City, UT, Salt Lake City, Utah, United States

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Result] Wambaugh JL, Wright S, Mauszycki SC, Nessler C, Bailey D. Combined aphasia and apraxia of speech treatment (CAAST): Systematic replications in the development of a novel treatment. Int J Speech Lang Pathol. 2018 Apr;20(2):247-261. doi: 10.1080/17549507.2016.1267262. Epub 2017 Jan 13. PMID 28084854
- [Result] Wambaugh JL, Wright S, Nessler C, Mauszycki SC. Combined Aphasia and Apraxia of Speech Treatment (CAAST): effects of a novel therapy. J Speech Lang Hear Res. 2014 Dec;57(6):2191-207. doi: 10.1044/2014_JSLHR-L-14-0004. PMID 25075917
- [Result] Bailey DJ, Blomgren M, DeLong C, Berggren K, Wambaugh JL. Quantification and Systematic Characterization of Stuttering-Like Disfluencies in Acquired Apraxia of Speech. Am J Speech Lang Pathol. 2017 Jun 22;26(2S):641-648. doi: 10.1044/2017_AJSLP-16-0108. PMID 28654945
- [Derived] Haley KL, Smith M, Wambaugh JL. Sound Distortion Errors in Aphasia With Apraxia of Speech. Am J Speech Lang Pathol. 2019 Feb 21;28(1):121-135. doi: 10.1044/2018_AJSLP-17-0186. PMID 31072155
- [Derived] Bunker LD, Nessler C, Wambaugh JL. Effect Size Benchmarks for Response Elaboration Training: A Meta-Analysis. Am J Speech Lang Pathol. 2019 Mar 11;28(1S):247-258. doi: 10.1044/2018_AJSLP-17-0152. PMID 30054623
- [Derived] Bunker LD, Wright S, Wambaugh JL. Language Changes Following Combined Aphasia and Apraxia of Speech Treatment. Am J Speech Lang Pathol. 2018 Mar 1;27(1S):323-335. doi: 10.1044/2018_AJSLP-16-0193. PMID 29497747

RESULTS

PARTICIPANT FLOW:
Groups:
- Combined Aphasia and Apraxia of Speech Treatment (CAAST): CAAST was administered to 4 persons with aphasia and apraxia of speech in the context of single-subject designs
  Combined Aphasia and Apraxia of Speech Treatment (CAAST): Therapy is delivered in a face-to-face format. The therapist uses picture stimuli, verbal modeling, feedback, reinforcement, forward-chaining to increase verbal production. For speech errors that occur, the therapist uses modeling, feedback, reinforcement, simultaneous production, articulatory instruction, and repeated practice to improve articulation.
Period: Overall Study
Arm/Group | Combined Aphasia and Apraxia of Speech Treatment (CAAST)
Started | 4
Completed | 4
Not Completed | 0

BASELINE CHARACTERISTICS:
Groups:
- Combined Aphasia and Apraxia of Speech Treatment (CAAST): Speakers with chronic aphasia and apraxia of speech who received the experimental treatment
Arm/Group | Combined Aphasia and Apraxia of Speech Treatment (CAAST)
Number analyzed (Participants) | 4
Age, Continuous [Mean (Full Range); unit: years] | 51 [39 to 69]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 2
  Male | 2
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 1
  Asian | 0
  Native Hawaiian or Other Pacific Islander | 0
  Black or African American | 0
  White | 3
  More than one race | 0
  Unknown or Not Reported | 0
Region of Enrollment [Count of Participants; unit: Participants]
  United States | 4

OUTCOME MEASURES:

1. Primary Outcome: Change in Language Content Production for Treated Stimuli: Effect Sizes (Magnitude of Change From Baseline to Follow-up)
Description: Correct Information Units (CIUs) is a measure of the amount of relevant content produced in connected language tallied according to operationalized criteria. CIU is not a test or scale - it is a measure that is applied to language samples - in this case, description of treated pictures. Participants described experimental pictures, responses were transcribed and CIUs counted. CIUs can range from 0 to an unlimited maximum. Effect sizes (ESs) were calculated as an indication of the magnitude of change in number of CIUs produced (pre treatment to post treatment. ESs can range from negative (poorer performance post-treatment) to positive values (better performance post-treatment), with larger positive values reflecting greater gains. Benchmarks are as follows: >11.14 = large, 11.13 - 6.56 = medium, 6.55 - 3.88 = small, <3.88 = negligible. Small to large ESs indicate production of measurably more CIUs in picture descriptions post-treatment. Larger the ES, the greater the change.
Time Frame: Following completion of treatment at 6 weeks post
Measure: Mean (Full Range); unit: units on a scale
Groups:
- Combined Aphasia and Apraxia of Speech Treatment (CAAST): CAAST was administered to 4 persons with aphasia and apraxia of speech in the context of single-subject designs.
Arm/Group | Combined Aphasia and Apraxia of Speech Treatment (CAAST)
Number analyzed (Participants) | 4
units on a scale | 13.38 [1.54 to 42.77]

2. Primary Outcome: Change in Production of Language Content for Untreated Sets - Generalization Measured in Effect Sizes
Description: Correct Information Units (CIUs) is a measure of the amount of relevant content produced in connected language tallied according to operationalized criteria. CIU is not a test or scale - it is a measure that is applied to language samples - in this case, description of untreated pictures. Participants described experimental pictures, responses were transcribed and CIUs counted. CIUs can range from 0 to an unlimited maximum. Effect sizes (ESs) were calculated as an indication of the magnitude of change in number of CIUs produced (pre treatment to post treatment. ESs can range from negative (poorer performance post-treatment) to positive values (better performance post-treatment), with larger positive values reflecting greater gains. Benchmarks are as follows: >9.53 = large, 9.52 - 5.52 = medium, 6.55 - 3.29 = small, <3.29 = negligible. Small to large ESs indicate production of measurably more CIUs in picture descriptions post-treatment. Larger the ES, the greater the change.
Time Frame: baseline (prior to treatment) through follow-up at 6 weeks post treatment
Population: One participant received treatment on all sets; consequently, generalization to an untreated set could not be calculated
Measure: Mean (Full Range); unit: units on a scale
Arm/Group | Combined Aphasia and Apraxia of Speech Treatment (CAAST)
Number analyzed (Participants) | 3
units on a scale | 7.99 [.89 to 15.54]

3. Secondary Outcome: Changes in Speech Intelligibility on the Assessment of Intelligibility of Dysarthric Speech
Description: Speech intelligibility (understandability of speech) was measured by having participants produce 50 words from the Assessment of Intelligibility of Dysarthric Speech (ASSIDS) Two speech-language (blinded) scored pre and post treatment ASSIDS samples. The percentage of words correctly understood was calculated for each participant. The ASSIDS is not a scale - it is a procedure for calculating intelligibility. Speech intelligibility can range from 0% to 100% intelligible (no words understood to all words understood). The higher the percentage, the better the speech is understood by the listener. Change in percent words intelligible has the potential to be a negative (reflecting a poor outcome of less intelligible speech) or positive (reflecting a good outcome of more intelligible speech). The maximum possible amount of gain in intelligibility for these 4 participants, based on their pretreatment performance, ranged from +2% to +25%.
Time Frame: pre and post treatment - prior to the start of treatment and at 6 weeks following the completion of treatment
Population: Change in percent of words that were intelligible
Measure: Mean (Full Range); unit: percentage of change-intelligible words
Groups:
- Combined Aphasia and Apraxia of Speech Treatment (CAAST): CAAST was administered to 4 persons with chronic aphasia and apraxia of speech in the context of single-subject designs
Arm/Group | Combined Aphasia and Apraxia of Speech Treatment (CAAST)
Number analyzed (Participants) | 4
percentage of change-intelligible words | 6.75 [0 to 10]

ADVERSE EVENTS:
Time Frame: Adverse event data were collected for the entire study duration for each participant: baseline/assessment period, treatment period, and through 6 week post-treatment period.
Groups:
- Combined Aphasia and Apraxia of Speech Treatment (CAAST): Administration of CAAST to 4 persons with aphasia and apraxia of speech in the context of single-subject designs
  Combined Aphasia and Apraxia of Speech Treatment (CAAST): Therapy is delivered in a face-to-face format. The therapist uses picture stimuli, verbal modeling, feedback, reinforcement, forward-chaining to increase verbal production. For speech errors that occur, the therapist uses modeling, feedback, reinforcement, simultaneous production, articulatory instruction, and repeated practice to improve articulation.
Arm/Group | Combined Aphasia and Apraxia of Speech Treatment (CAAST)
All-Cause Mortality (participants affected / at risk) | 0/4
Serious Adverse Events (participants affected / at risk) | 0/4
Other Adverse Events (participants affected / at risk) | 0/4

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No